CLINICAL TRIAL: NCT05926284
Title: Prospective Observational Study of a Precision Medicine Approach in Patients With Advanced Cancer
Acronym: PRIME
Status: Recruiting | Type: Observational
Sponsor: Charite University, Berlin, Germany (Other)
Responsible Party: Principal Investigator, Damian Rieke, Speaker, Platform for personalized cancer therapy at Charité Comprehensive Cancer Center, Principal Investigator, Medical Doctor, Charite University, Berlin, Germany
Other Study IDs: 3000764
Record Dates: First submitted 2023-04-08; First posted 2023-07-03 (Actual); Last update posted 2023-07-03 (Actual); Status verified 2023-06

CONDITIONS: Cancer
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Prospective observational study of a precision medicine approach in patients with advanced cancer. In this registrational study, patients with advanced cancer undergoing extensive molecular sequencing within the precision oncology program of Charité University Medicine, Berlin will be registered and followed to assess the efficacy of the program and assess the clinical relevance and frequency of molecular alterations, individualized therapies and novel molecular analysis tools.

ELIGIBILITY:
Inclusion Criteria:

* advanced cancer
* ability to give written informed consent
* performance status allows initiation of a potential targeted treatment after molecular analysis
* molecular analysis has been done or planned

Exclusion Criteria:

- unable to give written informed consent

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients with advanced cancer presenting to the precision oncology program at Charité for molecular analyses to identify personalized treatment options.
Sampling Method: Non-Probability Sample
Enrollment: 2000 (Estimated)
Dates: Start 2016-03-01 (Actual); Primary Completion 2030-03-01 (Estimated); Study Completion 2031-03-01 (Estimated)

PRIMARY OUTCOMES:
Frequency of personalized treatment initiation | At 1 year from date of study inclusion
  Frequency of personalized treatment initiation
Frequency of molecularly stratified treatment options | At 1 year from date of study inclusion
  Number of molecularly stratified treatment options per patient

SECONDARY OUTCOMES:
Progression free survival | Assessed up to 100 months
  From date of study inclusion until the date of first documented progression or date of death from any cause, whichever came first
PFS-ratio | Assessed up to 100 months
  Ratio of progression-free survival with molecularly matched therapy to progression-free survival with previous treatment line
objective response rate | 1 year after study inclusion
  Best radiographic response as assessed by the investigator
frequency of interventional study inclusion | At 1 year after study inclusion
  Number of participants with inclusion in interventional clinical trial
frequency of re-diagnosis | At 1 year after study inclusion
  Number of participants with a change in diagnosis a
frequency of recommendation of genetic counselling | At 1 year after study inclusion
  Number of participants with a recommendation for genetic counselling
frequency of pharmacogenomic findings | At 1 year after study inclusion
  Number of participants with a recommendation for pharmacongenomic considerations a
frequency and type of resistance mutations | At 1 year after study inclusion
  Number of molecular alterations predicting resistance to molecularly matched therapy a
overall survival | Assessed up to 100 months
  From date of study inclusion until the date of death from any cause, whichever came first
Evidence level of molecularly stratified treatment options | At 1 year from study inclusion
  Frequency of evidence levels (according to NCT evidence levels) of molecularly stratified treatment options

CONTACTS AND LOCATIONS:
Locations (1):
- Charité Comprehensive Cancer Center, Berlin, Germany